CLINICAL TRIAL: NCT01920828
Title: Gait Analysis in Patients With MPS IVA Treated With Enzyme Replacement Therapy
Brief Title: Gait Analysis in MPS IVA
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Utah (Other); BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: OregonHSU-8833
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: MPS IVA; Morquio Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to learn about gait (walking) characteristics in MPS IVA and possible changes in gait with enzyme replacement therapy.

DETAILED DESCRIPTION:
The purpose of this 3-year study is to conduct a longitudinal investigation using motion analysis of gait to objectively and quantitatively assess gait characteristics of MPS IVA patients. Data documenting gait characteristics and abnormalities will be gathered in patients initiating enzyme replacement therapy.

Inclusion criteria Individuals with MPS IVA diagnosed by enzyme or molecular studies Exclusion Criteria Individual with MPS IVA previously enrolled in BMN-110 Individual is non-ambulatory The individual is unable to complete longitudinal study visits at least yearly

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of MPS IVA

Exclusion Criteria:

Non-ambulatory

* Previous enrolled in clinical trial BMN-110

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of MPS IVA
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Measurable changes in gait | 36 months
  Data acquired on patients will be compared with age-matched standardized norms. The normal data is available from a pre-existing Gait Repository, a collection of gait parameters in children without a specific diagnosis studied at Oregon Health and Science University. The results will be converted to centile charts with the aid of a biostatistician. Centile charts will be used to track statistical changes over time in the following gait parameters including but not exclusive to: velocity, cadence, step length, and base of support.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States